CLINICAL TRIAL: NCT07011368
Title: Empowering Healthy Lifestyle Behaviour Through Personalized Intervention Portfolios to Prevent and Control Obesity During Vulnerable Stages of Life: The HealthyW8 Project.
Brief Title: Empowering Healthy Lifestyle Personalised Intervention to Prevent and Control Obesity: The HealthyW8 Project
Acronym: HealthyW8
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Collaborators: Luxembourg Institute of Health (Other Government); University of Évora (Other); University of Coimbra (Other); Eindhoven University of Technology (Other); Leibniz Institute for Prevention Research and Epidemiology - BIPS GmbH (Other); Deutsches Forschungszentrum für Künstliche Intelligenz (DFKI) (Unknown); Technical University of Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HealthyW8-Pilot-and-Long-Trial; 101080645 (Other: EU Horizon)
Record Dates: First submitted 2025-04-07; First posted 2025-06-08 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-04

CONDITIONS: Obesity Prevention; Obesity and Overweight; Obesity and Obesity-related Medical Conditions; Digital Health; Behavioural Science Interventions to Improve Health Equity
Keywords: Healthy lifestyle recommender system; digital empowerment; health literacy; personalised prevention; pre-obesity biomarkers; mHealth; Human Digital Twin; behavior change techniques; physical activity
MeSH Terms: conditions — Obesity; Overweight; Motor Activity

STUDY DESIGN:
Intervention Model Description: Intervention:
  1. Pilot studies: Main objective is to validate the selected tool-assisted interventions by iteratively testing the HLRS and other health intervention tools among different end-user groups within different contexts (e.g. cultural, economic, social, physical). Pilot trials (<3 months; n=30 per each age group: children, young adults, and elders) will assess their efficacy considering psychological/emotional states, adherence to dietary suggestions, technology acceptance, efficacy of nudges/gamification, user-friendliness of the tools, and actual usage and engagement. Outcomes will provide feedback for HLRS, including input for the HDT, and a roadmap for long-term intervention studies.
  2. Long-trials: Main objective is to assess the effect of 1-y interventions with the HLRS described and further iteratively improved in Pilot trial on reducing risk of overweight/obesity at described life-stages n=55 per control & intervention group, and described ages).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- School-children (including families) (Experimental): HLRS intervention on 5-12 year-old school-children (including families) adapted to the countries in which they will be deployed (e.g.: adaptation to cultural food habits, translation into national languages).
  Interventions: Behavioral: Intervention Group
- Young adults (Experimental): HLRS intervention on 18-25-year-old young adults adapted to the countries in which they will be deployed (e.g.: adaptation to cultural food habits, translation into national languages).
  Interventions: Behavioral: Intervention Group
- Elderly people (Experimental): HLRS intervention on >65-year-old elderly people adapted to the countries in which they will be deployed (e.g.: adaptation to cultural food habits, translation into national languages).
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — Healthy Lifestyle Recommender Solution (HLRS) will be developed as intervention tool for the trials. It integrates tools (mostly digital): a meal recommender to propose balanced and individually adapted meal plans, physical activity and sleep pattern measures and recommendations, assessment of behavioural/psychological aspects, and motivational features for sustained engagement and adherence.
  Within our multi-disciplinary portfolio approach, a set of predominantly eHealth solutions applied during the intervention trials for overweight/obesity prevention, developed in a participatory design approach with relevant stakeholders. This will include the HLRS, thus combining motivational features (nudging, gamification), targeted psychological support, dietary and physical activity advice, though also additional recommendations (healthy eating guidelines...) or education materials will be provided.
  Intervention trials/studies.

SUMMARY:
The goal of the HealthyW8 study (an intervention study) is:

To assess the usefulness and effects of a digital-based healthy lifestyle recommender system (HRLS) on the prevention of obesity in the following propulations: schoolchildren (5-10 y) and their parents, young adults (18-25 y) and elders (>65 y).

The main questions it aims to answer are:

Outcome 1: To select and validate a tool-assisted 3-mo intervention (mostly digital) by iteratively testing the HLRS on reducing risk of overweight/obesity among the described age groups.

Outcome 2: To assess the effect of 1-y interventions (mostly digital) with the HLRS described and further iteratively improved previously (outcome 1) on reducing risk of overweight/obesity at described ages.

Researchers will compare the intervention group before the intervention (baseline) and after it (3-mo intervention trial), or control group (standard care) vs. Intervention group (1-y intervention) to see changes on changes in overweight/obesity, and related parameters (body composition and biomarkers).

Participants will follow the HLRS recommendations (meal plans, physical activity and sleep pattern measures and recommendations, assessment of behavioural/psychological aspects, and motivational features through digital devices), which will be assessed by means of measurement of body weight, body composition, and biomarkers.

DETAILED DESCRIPTION:
HealthyW8 will enhance early screening and prevention of obesity by making the scientific and technological breakthroughs necessary to support evidence-based clinical, environmental and policy-level decisions, while also directly empowering citizens to adopt healthy and sustainable lifestyle behaviours in a "push-pull" approach.

HealthyW8 will step up primary obesity prevention efforts across Europe, endowing them with a multi-disciplinary portfolio approach, i.e. a set of selective multi-component interventions that combine a large set of interventions and implementation options, focussing on diet, physical activity (PA), and psycho-emotional aspects.

The current approach considers obesity as a multifactorial phenomenon, necessitating a holistic, systemic approach accounting for the complexity of individual, interpersonal, organisational, community and public policy levels, as mutually reinforcing and supportive systems.

The attention will be focused on pivotal situations of transitions in the life-trajectory of individuals, which pose an elevated risk to progress from healthy weight to overweight and obesity, i.e. windows of opportunity to reduce the risk of developing obesity where the impact will have most leverage.

HealthyW8 targets vulnerable populations where transitional changes of lifestyle appear to be dominant: primary schoolchildren (5-12y, with active parent involvement), young adults (18-25y), and the elderly (>65y).

A central pillar of the current multiportfolio approach and intervention strategy will be a healthy lifestyle recommender solution (HLRS). Despite many apps on the market today that propose changes in dietary behaviour/PA, overweight and obesity are still on the rise across Europe. They failed to engage citizens with low interest in healthy lifestyle patterns and suffer from prominent limitations that HealthyW8 will address by developing the HLRS as a core element of our adapted intervention strategy and appropriate intervention tools.

Interventions' acceptability and feasibility to key stakeholders will be ensured by a participatory design approach, allowing stakeholders to influence from the outset their design & development and integrate the needs of the target groups. The obesity prevention potential of interventions and/or their implementation strategies will be evaluated in over a dozen multicentre pilots (<3 months) and long-term (12 months) randomised control trials (RCTs). In parallel, it will collect user feedback on feasibility, acceptability and needs, allowing researchers to respond in real-time to problems/deviations and to capture context-related factors of success/failure.

Applying SMART criteria, HealthyW8 will achieve the following objectives:

1. Expand understanding of the biological causes underlying obesogenic trends & interactions with crosscutting environmental, behavioural & policy factors to propose evidence-based effective obesity prevention strategies.
2. Develop user-centred portfolio interventions to enhance the impact on lifestyle changes in an efficient, synergistic, long-lasting & sustainable way.
3. Iteratively optimise the intervention strategies involving vulnerable populations/those undergoing transitions to maximise impact.
4. Leverage findings to EU stakeholders & foster the multilevel uptake of solutions & strategies.

Accordingly, multi-disciplinary portfolios of interventions adaptable to the targeted populations, and further to the individual (anthropometry, general health aspects, inflammation, oxidative stress, epigenetics, omics, microbiota, dietary & general consulting, healthy lifestyle recommender solutions - HLRS, Human Digital Twin - HDT, policies recommendations, Open Stakeholder Pltform - OSP) will be developed. The focus on primary prevention, specifically the progression from healthy weight to overweight/obese, will allow targeting a broader population with a better cost/benefit ratio than secondary/tertiary preventions, though anticipating that the current portfolio approach and HLRS are adaptable to treatment scenarios also.

After an inventory of best practises & relevant levers for overweight/obesity prevention & management existing literature evidence will be synthesised. A system map for obesity prevention for the different targeted vulnerable groups and for the HDT. Via scoping, systematic and (umbrella-) reviews/meta-analyses, main drivers of the obesogenic environment will be highlighted.

These findings will be integrated in a multi-actor participatory design approach (Design Thinking, DT) into the development of the HLRS and of the HDT.

Implementation of pilot trials (<3 month; n=30 for each age group: primary schoolchildren (5-12y, with active parent involvement), young adults (18-25y), and the elderly (>65y) will be applied to validate the selected tool-assisted interventions by testing the HLRS and other health intervention strategies & tools. Outcomes will lead to iterative tool development and a roadmap for larger long-term intervention studies.

Long term RCTs (12 months) with the same population groups will be conducted (n=55 per age group), compared vs. controls (n=55 per age group; receiving standard recommendations).

Populations will be replicated several times, participants longitudinally followed, and outcomes collected including: a) eating patterns (FFQs); b) markers related to obesity and comorbidities; c) lifestyle and cognitive aspects, psycho-emotional well-being (Emotional Guidance Scale encompassing e.g. joy, appreciation, freedom, empowerment, despair, fear); d) technological acceptance and usability (Mobile Application Rating Scale). Hence, we will apply a biopsychosocial understanding of obesity, integrating physiological, psychosocial, and contextual factors into one coherent model. Many markers/measures will be identical between countries/populations (core-endpoints), some different due to local/population-required adaptations.

Main outcome will be to assess the effect of 1 y interventions with the HLRS described and further iteratively improved in Pilot studies on reducing risk of overweight/obesity at various life-stages. Secondary objectives will be to assess the effect of interventions on body composition and metabolic and other parameters.

ELIGIBILITY:
Inclusion Criteria:

* Overweight (BMI between 25-30 kg/m^2)
* To have a smart phone

Exclusion Criteria:

* Individuals with manifest chronic diseases
* Individuals with cognitive diseases
* Individuas not able to lead an independent life

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2720 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in BMI | Baseline and every 3 months up to 12 months
  The Primary Outcome (to be measured every 3 months) will be the change of BMI (kg/m^2) measuring body weight in kilograms and height in meters^2 as combined to obtain BMI data (kg/m^2) after the 12-month intervention of healthy lifestyle recommender solutions (HLRS) in the selected age groups (5-12 y.o. children and families; 18-25 y.o. young adults; and >65 y.o. elderly people).

SECONDARY OUTCOMES:
Change of visceral body fat | Baseline and every 3 months up to 12 months
  The Secondary Outcome (to be measured every 3 months) will be the change of visceral body fat measuring body fat in kilograms and in percentage of body weight after the 12-month intervention of healthy lifestyle recommender solutions (HLRS) in the selected age groups (5-12 y.o. children and families; 18-25 y.o. young adults; and >65 y.o. elderly people).
Body composition and biomarkers | Baseline and every 6 months up to 12 months
  Other Secondary outcomes will be several biological markers measured every 6 months:
  * lipidic profile (cholesterol, LDL-c, HDL-C, triglycerides): mg/dL
  * glycidic profile (fasting blood glucose, HbA1C, insulin): mg/dL
  * inflammatory biomarkers (CRP, IL-1b/6/8, TNFa)
  * oxidative stress biomarkers (F2-isoprostanes, malondialdehyde): ng/mL
  * nutrition related markers: vitamin E, total carotenoids, total phenolics, sodium in urine: ng/dL
  * gut microbiome analyses (16S rRNA): assessment of bacterial species

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Bohn, PhD, Principal Investigator — Luxembourg Institute of Health
Locations (13):
- Bulgaria (2):
  - Virtech Ood, Sofia
  - Regional Cluster North-East, Varna
- Danmarks Tekniske Universitet, Kongens Lyngby, Denmark
- Germany (2):
  - Leibniz-Institut Fur Praventionsforschung Und Epidemiologie - Bips Gmbh, Bremen
  - Deutsches Forschungszentrum Fur Kunstliche Intelligenz Gmbh, Kaiserslautern
- Universita Degli Studi Di Scienze Gastronomiche, Bra, Italy
- Luxembourg Institute of Health, Luxembourg, Luxembourg
- Technische Universiteit Eindhoven, Eindhoven, Netherlands
- Portugal (2):
  - Universidade de Coimbra, Coimbra
  - Universidade de Evora, Evora
- Spain (3):
  - Fundacio Institut D'Investigacio Sanitaria Illes Balears (Idisba), Palma de Mallorca, Balearic Islands
  - Centre de Recerca En Economia I Desenvolupament Agroalimentari-Upc-Irta, Castelldefels
  - Centro de Investigacion Y Tecnologia Agroalimentaria de Aragon, Zaragoza

IPD SHARING:
Plan to Share IPD: No
There are restrictions on the availability of data for this trial, due to the signed consent agreements around data sharing, which only allow access to external re-searchers for studies following the project purposes. Researchers wishing to access the trial data used in this study can make a request to pep.tur@uib.es

REFERENCES:
- [Background] Vahid F, Dessenne C, Tur JA, Bouzas C, Devaux Y, Malisoux L, Monserrat-Mesquida M, Sureda A, Desai MS, Turner JD, Lamy E, Perez-Jimenez M, Ravn-Haren G, Andersen R, Forberger S, Nagrani R, Ouzzahra Y, Fontefrancesco MF, Onorati MG, Bonetti GG, de-Magistris T, Bohn T. Multicomponent (bio)markers for obesity risk prediction: a scoping review protocol. BMJ Open. 2024 Mar 8;14(3):e083558. doi: 10.1136/bmjopen-2023-083558. PMID 38458803
- See also: HealthyW8: Empowering Healthy Lifestyle Behaviour — https://www.healthyw8.eu/